CLINICAL TRIAL: NCT02616757
Title: Quantitative Ultrasound for the Evaluation of Simple Bone Cyst Healing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Ultrasound machine was no longer approved for use by Health Canada therefore study was closed prior to patients being enrolled on study.
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, James Wright, Orthopaedic Surgeon, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000049774
Record Dates: First submitted 2015-11-25; First posted 2015-11-30 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Simple Bone Cyst
MeSH Terms: conditions — Bone Cysts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Simple Bone Cyst Patients (Active Comparator): Z-score measurements will be taken from the mid-shaft tibia and distal third of the radius of both extremities where possible using quantitative ultrasound at baseline and once annually for 2 years.
  There will also be optional blood samples taken o measure bone alkaline phosphatase.
  Interventions: Device: Sunlight Omnisense Quantitative Ultrasound
- Fracture patients (Active Comparator): Z-score measurements will be taken from the mid-shaft tibia and distal third of the radius of both extremities where possible using quantitative ultrasound at baseline, after 3 months and at future follow-up visits as clinically indicated or at a one year follow-up visit.
  There will also be optional blood samples taken to measure bone alkaline phosphatase.
  Interventions: Device: Sunlight Omnisense Quantitative Ultrasound
- Health volunteers (Placebo Comparator): Z-score measurements will be taken from the mid-shaft tibia and distal third of the radius of both extremities where possible using quantitative ultrasound at baseline, after 3 months and at a one year follow-up visit.
  There will also be optional blood samples taken to measure bone alkaline phosphatase.
  Interventions: Device: Sunlight Omnisense Quantitative Ultrasound

INTERVENTIONS:
Device: Sunlight Omnisense Quantitative Ultrasound — Ultrasound

SUMMARY:
Simple bone cysts (SBCs), also known as unicameral bone cysts (UBCs), are benign bone lesions. Literature to date describes little agreement between clinicians on specific prognostic criteria for the prediction of cyst healing, recurrence or fracture. Evidence has shown that bone mineral density (BMD) is a reliable indicator of risk to SBC patients given its association with the mechanical properties of bone. There has been further exploration into the use of quantitative ultrasound to assess bone density by measuring the velocity of the ultrasound transmission over the bone. To determine whether the QUS can provide prognostic information with respect to cyst healing, recurrence or fracture with a SBC, further study is needed.

ELIGIBILITY:
Arm 1 - Simple Bone Cyst Patients

Inclusion Criteria

1. Patients ≥ 2 and ≤ 21 years
2. Patients with a diagnosis of simple bone cyst located in a long bone confirmed by imaging within 3 months prior to registration
3. All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria

1. Patients with implants to stabilize the bone where the cyst is located.
2. Patients with bone disease (i.e. osteogenesis imperfecta, cancer, osteoporosis, Paget's disease)
3. Patients who are pregnant or breastfeeding
4. Patients with a simple bone cyst crossing the growth plate

Arm 2 - Healthy Controls

Inclusion Criteria

1. Patients ≥ 2 and ≤ 21 years
2. All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria

1. Patients with bone disease (i.e. osteogenesis imperfecta, cancer, osteoporosis, Paget's disease)
2. Patients receiving any bone-modifying agents (i.e. steroids, bisphosphanates, etc.)
3. Patients who are pregnant or breastfeeding

Arm 3 - Fracture patients

Inclusion Criteria

1. Patients ≥ 2 and ≤ 21 years
2. Patients who have undergone any type of casting or surgical treatment for their fracture
3. All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria

1. Patients with bone disease (i.e. osteogenesis imperfecta, cancer, osteoporosis, Paget's disease)
2. Patients receiving any bone-modifying agents (i.e. steroids, bisphosphanates, etc.)
3. Patients who are pregnant or breastfeeding

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-06 (Actual)

PRIMARY OUTCOMES:
Z-scores obtained using quantitative ultrasound | 2 years

SECONDARY OUTCOMES:
Bone specific alkaline phosphatase | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Howard, MD, Principal Investigator — The Hospital for Sick Children; James G. Wright, MD, Principal Investigator — Nuffield Orthopaedic Centre
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada